CLINICAL TRIAL: NCT04387916
Title: A Phase I, Open-label, Dose Escalation Study Evaluating the Safety, Pharmacokinetics and Preliminary Efficacy of KC1036 in the Patients with Advanced Recurrent or Metastatic Solid Tumors
Brief Title: A Study of KC1036 in Patients with Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Konruns Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KC1036-I-01
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- KC1036 (Experimental): Patients take a single dose of KC1036 for the pharmacokinetic study, then off for 5 days before the first cycle begins. In the subsequent treatment cycles, KC1036 are given orally once daily, 21 days as a cycle.
  Interventions: Drug: KC1036

INTERVENTIONS:
Drug: KC1036 — Part 1: Dose-escalation phase , KC1036 10mg~80mg, consists of 5 Cohorts. Part 2: Dose-expansion phase, consists of 3~4 Cohorts based on part 1. Part 3:RP2D-extension phase, Recommended dose of KC1036 based on part 1and part 2.

SUMMARY:
The purpose of this study is to evaluate the safety，tolerability, pharmacokinetics, and preliminary efficacy of KC1036 in participants with advanced recurrent or metastatic solid tumors. The trial will be divided into three parts: dose-escalation phase, dose-expansion phase, RP2D-extension phase.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed recurrent or metastatic solid tumors;
* Patients who have failed standard or conventional treatment, Including chemotherapy, targeted therapy, immunotherapy:

Documented disease progression after, or refractory to, or intolerant of prior standard or established therapy known to provide clinical benefit for their condition; or documented disease progression within 24 weeks after prior adjuvant/neoadjuvant therapy;

* At least one measurable lesion (by RECIST 1.1);
* Eastern Cooperative Oncology Group performance status score of 0 or 1;
* Life expectancy > 12 weeks;
* Patients should participate in the study voluntarily and sign informed consent.

Exclusion Criteria:

* Untreated brain metastases or symptoms of brain metastases cannot be controlled more than 4 weeks;
* Other kinds of malignancies;
* Hematologic, renal, and hepatic function abnormities;
* Risk of bleeding;
* Gastrointestinal abnormalitiest;
* Cardiovascular and cerebrovascular diseases;
* Prior anti-tumor therapies with chemotherapy, radiotherapy, hormonotherapy, biotherapy, immunotherapy, operation within 4 weeks of enrollment;
* Presence of unresolved toxicities from prior anti-tumor therapy, defined as having not resolved to NCI CTCAE V5.0 grade 0 or 1 with the exception of alopecia;
* Involved in other clinical trials within 4 weeks of enrollment;
* Major surgical procedure, open biopsy, or significant traumatic injury 4 weeks days of enrollment;
* History of organ allograft;
* Need immunosuppressive agents or systemic or absorbable topical hormone therapy for immunosuppression;
* Uncontrolled ongoing or active infection;
* Known history of human immunodeficiency virus (HIV) infection or current chronic or active hepatitis B or C infection requiring treatment with antiviral therapy;
* Pregnant or lactating women or those who do not take contraceptives, including men;
* Suffering from mental and neurological diseases;
* Any other metabolic dysfunction, abnormal physical examination findings, or clinical laboratory findings;
* Inability to comply with protocol required procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Estimated)
Dates: Start 2020-09-04 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | First 4 weeks after initial administration of KC1036
  MTD will be defined as the maximum dose level at which no more than 1 of 3 participants experience a dose-limiting toxicity (DLT) within the first 4 weeks of multiple dosing.
Adverse events (AEs) | From enrollment up to 30 days after last dose
  Incidence of treatment-related AEs

SECONDARY OUTCOMES:
Pharmacokinetics (PK) profile: Cmax | First 4 weeks after initial administration of KC1036
  Peak Plasma Concentration
Pharmacokinetics (PK) profile: Tmax | First 4 weeks after initial administration of KC1036
  Time to reach the maximum plasma concentration
Pharmacokinetics (PK) profile: T1/2 | First 4 weeks after initial administration of KC1036
  Terminal half-life
Pharmacokinetics (PK) profile: AUC0-t and AUC0-∞ | First 4 weeks after initial administration of KC1036
  Area under the single-dose plasma concentration-time curve from Hour 0 to the last quantifiable measurable plasma concentration, or Area under the single-dose plasma concentration-time curve from Hour 0 to infinity
Objective Response Rate (ORR) | Every 6 weeks for the duration of study participation; estimated to be 12 months
  Overall response rate (ORR) was defined as the percentage of participants with a best overall complete response (CR) or partial response (PR) per RECIST 1.1.
Progression-free survival (PFS) | Every 6 weeks for the duration of study participation; estimated to be 12 months
  Progression-free survival (PFS) was defined as the time from the start date of study drug to the date of the first radiologically documented progressive disease (PD) per RECIST 1.1 or death due to any cause.
Disease Control Rate (DCR) | Every 6 weeks for the duration of study participation; estimated to be 12 months
  Disease Control Rate (DCR) was defined as the percentage of participants with a best overall complete response (CR), partial response (PR), or stable disease (SD) per RECIST 1.1.
Duration of Response (DOR) | Every 6 weeks for the duration of study participation; estimated to be 12 months
  Duration of response (DOR) was defined as the time from first documented response (partial response (PR) or complete response (CR)) to the date of first documented disease progression (PD) or death due to any cause, among patients with a confirmed PR or CR per RECIST 1.1.
Overall Survival (OS) | From the first medication to death due to any cause; estimated to be the subject's death, loss to follow-up, or end of the study]
  Overall Survival (OS) was defined as the time from the start date of study drug to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - ChongQing University Cancer Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - West China Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No